CLINICAL TRIAL: NCT05903443
Title: Research on the Brain Death Determination and Quality Controlin Chinese Adults
Brief Title: Research on the Brain Death Determination in China
Acronym: RBDDC
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2014004
Record Dates: First submitted 2023-05-24; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Brain Death; Electroencephalogram; Evoked Potential; TCD; Quality Control
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BD group: All cases met the (brain death) BD clinical evaluation criteria, which were as follows: the cause of coma was known; exclusion of reversible coma; deep coma, Glasgow coma scale (GCS) = 2T; absence of five brain stem reflexes (pupillary light reflex, corneal reflex, oculocephalogyric reflex, oculovestibular reflex, and cough reflex); and no spontaneous respiration. Furthermore, according to whether the apnea test (AT) data were missing (implemented or completed), the patients were divided into the BD1 group (no AT missing group) and BD2 group (AT missing group).
  Interventions: Diagnostic Test: ancillary tests
- non-BD group: All cases were from BDQCHs and fulfilled the criteria for coma (GCS of 3-5 points), but did not meet the clinical criteria for BD, such as retaining the brainstem reflex or having spontaneous respiration. For coma cases, all assessment items, specifications of technical operations, assessment steps, and evaluators were conducted in accordance with the requirements for BDD. Cases with coma were then submitted to the BQCC/NHC quality control system.
  Interventions: Diagnostic Test: ancillary tests

INTERVENTIONS:
Diagnostic Test: ancillary tests — electroencephalogram, short latency somatosensory evoked potential, transcranial Doppler

SUMMARY:
Purpose China has a population of 1.4 billion and an enormous medical expenditure burden, and Chinese traditional culture has a long history. It takes time to recognize and accept the concept of brain death (BD) as death. Promoting brain death determination (BDD) and rationally allocating medical resources have become major national policy issues. To identify the safest and most reliable ancillary tests needed if the clinical examination is incomplete.

Method The technical group of the Brain Injury Evaluation Quality Control Center of the National Health Commission retrieved coma cases registered from 2013 to 2019. According to clinical criteria for Brain Death Determination (BDD), the patients were divided into two groups: a brain-death (BD) group and a non-BD group. The BD group was divided into a complete brain death with no doubt group (BD1 group) and an incomplete brain death with doubt group (BD2 group). Depending on the site of the brain injury, the accuracy of BDD was evaluated using the independent ancillary test or combined ancillary tests. Data from the BQCC/NHC database and yearbook were obtained, and data analysis and status comparison were conducted on six practical activities: organizational system construction, standard and specification formulation, case quality control, professional skills training, scientific research publicity and education, and international communication.

ELIGIBILITY:
Inclusion Criteria:

* All cases met the clinical criteria for BD, involving deep coma (Glasgow Coma Scale (GCS)=2T), the absence of brainstem reflexes (pupillary light reflex, corneal reflex, oculocephalogyric reflex, oculovestibular reflex, and cough reflex), and spontaneous respiration. Ancillary tests were completed for all patients.

Exclusion Criteria:

* Does not meet BD clinical evaluation criteria. Ancillary tests were not implemented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coma cases registered by the National Brain Death Determination Quality Control Demonstration Hospital (BDQCH) in the BQCC/NHC from 2013 to 2019 were retrieved.
Sampling Method: Non-Probability Sample
Enrollment: 1974 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
sensitivity | 1 month
  The sensitivity of BDD was evaluated using the independent ancillary test and combined ancillary tests
specificity | 1 month
  The specificity of BDD was evaluated using the independent ancillary test and combined ancillary tests

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No